CLINICAL TRIAL: NCT02640768
Title: Governance of Diabetes Management in Non-specialistic Hospital Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Ivana Zavaroni, Associate Professor, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AOParma
Record Dates: First submitted 2015-11-19; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes
Keywords: in-hospital diabetes; clinical and management model
MeSH Terms: conditions — Diabetes Mellitus | interventions — Training Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- educational training (Experimental): educational training
  Interventions: Other: educational training
- no educational training (No Intervention): no educational training wards

INTERVENTIONS:
Other: educational training — implementation of a structured educational program for physicians and nurses
  Arms: educational training

SUMMARY:
The prevalence of diabetes among inpatients in medical wards, surgery and intensive care units in Italy is approximatively 12-25%. The management of in hospital diabetes and hyperglycemia is complex and requires a specific training for physicians and nurses in non-specialist settings. The overall project aims at the implementation of a "best practice" model of care for hospitalized diabetic patients in non-specialist settings.

DETAILED DESCRIPTION:
The project aims at defining a model of care for hospitalized diabetic patients in non-specialist settings based on the national and international recommendations. This is a cluster randomized study to evaluate the efficacy of a structured education training program for physicians and nurses in improving an ad hoc composite performance score of diabetes management and some clinical outcomes. The study will be carried out in 6 hospitals of the Emilia-Romagna region in Italy and it will involve 3 different wards (internal medicine, intensive care unit, surgery). For each hospital one intervention and two controls wards will be randomly identified.

At baseline the clinical management of patients with stress hyperglycemia/diabetes will be assessed in all participating wards over a 3-month period. Then, a structured educational program regarding the management of stress hyperglycemia/diabetes in the inpatient setting will be carried out only in the intervention wards. This program will last 2 months. Health care professionals also will be trained in the regular use of appropriate management tools (hyperglycemia dedicated standard operation procedures, audits, etc.).

Three months after the end of the educational program, the 3-month assessment of clinical management of patients with stress hyperglycemia/diabetes will be repeated in all participating wards.

The assessment of clinical management of stress hyperglycemia/diabetes will be based on a set of clinical performance indicators concerning 5 major domains (admission assessment, glucose monitoring, medical therapy, management of consults, management of discharge). These indicators will be used to define a composite performance score of appropriateness and efficacy. The highest score (1) will be assigned when the indicator is monitored, the lowest (0) when the indicator will be not detected, according to the scoring method previously reported by Rossi et al. Therefore, the score of each domain will range between 0 and the number of indicators used to assess appropriateness and efficacy of that domain.

Domain 1 - Initial assessment: score 0-5

* records of admission glycemia
* records of fasting plasma glucose
* records of HbA1c
* appropriate diagnosis of stress hyperglycemia/diabetes mellitus according to ADA
* records of history of presence/absence of pharmacological diabetes therapy

Domain 2 - Glucose monitoring: score 0-4

* appropriate glucose monitoring: at least 80% of three daily preprandial glycemia or, in critically ill patients, monitoring according to the specific algorithm used in the ward
* presence and use of specific forms for glucose records
* presence of ward standing orders to recognize and correct hypoglycemia
* presence of ward standing orders to monitor and manage glucose in critically ill patients (Critically ill patients are defined as patients who require intensive care for acute critical illnesses, such as myocardial infarction, stroke, septic shock or severe respiratory failure, requiring intensive or semi-intensive therapy and, as a rule, not taking food orally during the first 24-72 hours)

Domain 3 - Medical therapy: score 0-2

* records of time and dose of insulin therapy
* interruption of Metformin therapy when indicated (correct indications to discontinuation of Metformin therapy were: any critical illness, acute renal, cardiac and/or respiratory failure, surgery or iodinated contrast agents administration.)

Domain 4 - Consults: score 0-2

* request and records of diabetes specialist consult
* request and records of nursing consult

Domain 5 - Management of discharge: score 0-3

* planning of diabetes follow-up visit after hospitalization
* patient education for home blood glucose self-monitoring
* patient education for all other aspects of diabetes management

The sum of the scores of each domain from 1 to 5 is the composite performance score.

The following clinical outcomes will be recorded both at baseline and 3 months after the end of the educational program in all participating wards.:

* all hypoglycemic events (blood glucose ≤ 70 mg/dl)
* severe hypoglycemic events (blood glucose ≤ 40 mg/dl with or without clouding of consciousness)
* difference between plasma glycemia at admission and mean plasma glucose during the last-48-hours before discharge
* achievement of glycemic goals: 4 consecutive blood glucose levels ≤ 130 mg/dl (preprandial) or ≤ 180 mg/dl (postprandial), or 4 consecutive blood glucose levels between 140 and 180 mg/dl in critically ill patients
* survival
* discharge condition: a score of 0 will be assigned in case of death or transfer to a higher intensity ward and score 1 in all other cases, i.e. home discharge or transferral to a lower intensity ward.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 or type 1 diabetes or stress hyperglycemia

Exclusion Criteria:

* age <18,
* patients hospitalized for diabetic complications: ketoacidosis, hyperosmolar syndrome, hypoglycemic coma, pregnant diabetics or gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1449 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Composite performance score computed as the sum of the performance scores of all 5 domains of appropriateness and efficacy in both the intervention and the control wards | 11 months
  Efficacy of educational training will be evaluated as absolute change of the performance scores after the intervention compared to baseline in the two groups

SECONDARY OUTCOMES:
hypoglycemic events in the intervention and control wards | 11 months
  rate difference of hypoglycemia events (blood glucose ≤ 70 mg/dl) in the intervention and control wards
severe hypoglycemic events in the intervention and control wards | 11 months
  rate difference of severe hypoglycemia events (blood glucose ≤ 40 mg/dL with or without clouding of consciousness) in the intervention and control wards
difference between plasma glycemia at admission and mean plasma glucose during the last-48-hours before discharge | 11 months
  difference between plasma glycemia at admission and mean plasma glucose during the last-48-hours before discharge
achievement of glycemic goals in the intervention and control wards | 11 months
  number of patients that achieve glycemic goals: 4 consecutive blood glucose levels ≤ 130 mg/dl (preprandial) or ≤ 180 mg/dl (postprandial), or 4 consecutive blood glucose levels between 140 and 180 mg/dl in critically ill patients
survival rate during hospitalization in the intervention and control wards | 11 months
  survival rate during hospitalization (score 1 for survival, score 0 for death)
discharge condition in the intervention and control wards | 11 months
  a score of 0 will be assigned in case of death or transfer to a higher intensity ward and score 1 in all other cases, i.e. home discharge or transferral to a lower intensity ward.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Zavaroni, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Parma
Locations (6):
- Italy (6):
  - AUSL Ospedale Maggiore, Bologna
  - Azienda Ospedaliero-Universitaria, Ferrara
  - AUSL Carpi, Modena
  - Azienda Ospedaliero-Universitaria Parma, Parma
  - AUSL Piacenza, Piacenza
  - AUSL Montecchio, Reggio Emilia

REFERENCES:
- [Result] Cook CB, Castro JC, Schmidt RE, Gauthier SM, Whitaker MD, Roust LR, Argueta R, Hull BP, Zimmerman RS. Diabetes care in hospitalized noncritically ill patients: More evidence for clinical inertia and negative therapeutic momentum. J Hosp Med. 2007 Jul;2(4):203-11. doi: 10.1002/jhm.188. PMID 17683100
- [Result] Van den Berghe G, Wilmer A, Hermans G, Meersseman W, Wouters PJ, Milants I, Van Wijngaerden E, Bobbaers H, Bouillon R. Intensive insulin therapy in the medical ICU. N Engl J Med. 2006 Feb 2;354(5):449-61. doi: 10.1056/NEJMoa052521. PMID 16452557
- [Result] American Diabetes Association. Standards of medical care in diabetes--2008. Diabetes Care. 2008 Jan;31 Suppl 1:S12-54. doi: 10.2337/dc08-S012. No abstract available. PMID 18165335
- [Result] Rossi MC, Lucisano G, Comaschi M, Coscelli C, Cucinotta D, Di Blasi P, Bader G, Pellegrini F, Valentini U, Vespasiani G, Nicolucci A; AMD-QUASAR Study Group. Quality of diabetes care predicts the development of cardiovascular events: results of the AMD-QUASAR study. Diabetes Care. 2011 Feb;34(2):347-52. doi: 10.2337/dc10-1709. PMID 21270192